CLINICAL TRIAL: NCT03305250
Title: Arrhythmia Burden, Risk of Sudden Cardiac Death and Stroke in Patients With Fabry Disease: the Role of Implantable Loop Recorders
Brief Title: Arrhythmia Burden, Risk of Sudden Cardiac Death and Stroke in Patients With Fabry Disease
Acronym: RaILRoAD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Birmingham NHS Foundation Trust (Other)
Collaborators: Royal Free Hospital NHS Foundation Trust (Other); Northern Care Alliance NHS Foundation Trust (Other); University of Sydney (Other); Cambridge University Hospitals NHS Foundation Trust (Other); Cardiff and Vale University Health Board (Other Government); Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Dr Richard Steeds, Consultant in Cardiology, University Hospital Birmingham NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: FD-ILR-001
Record Dates: First submitted 2017-09-21; First posted 2017-10-09 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2024-12

CONDITIONS: Fabry Disease
MeSH Terms: conditions — Fabry Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Interventional Arm (Active Comparator): Using an Implantable Loop Recorder fo continuous rhythm monitoring and home follow-up. This will be combined with standard care procedure, which will include annual ECG, 24 hour Holter/5 day ECG monitoring and further investigation dependent on symptom status.
  Interventions: Device: Implantable Loop Recorder
- Standard of Care Arm (No Intervention): The standard of care with annual ECG, 24 hour Holter/5 day ECG monitoring and further investigation dependent on symptom status.

INTERVENTIONS:
Device: Implantable Loop Recorder — An implantable loop recorder (ILR), also known as an insertable cardiac monitor, is a small device (smaller than a AAA battery) that is inserted under the skin on the front of the chest. The ILR is inserted using local anesthetic as an out-patient procedure and lasts approximately 30 minutes. The ILR captures a continuous ECG of your heart activity, which allows doctors to detect any abnormal heart rhythms at any point. If you have the ILR, you will have the device for 3 years, after which it will be removed under local anesthetic during an out-patient procedure, again lasting approximately 30 minutes. The ILR device is completely safe and shouldn't affect your day to day living.
  Arms: Interventional Arm

SUMMARY:
Fabry disease (FD) is a genetic disorder that leads to progressive accumulation of fat or 'sphingolipid' within the tissues, including the heart muscle and conductive tissue. Improvements in the detection of FD, together with more organised clinical services for rare diseases, has led to a rapid growth in the disease prevalence. Earlier and more frequent diagnosis of asymptomatic individuals before development of the disease itself has focused attention on early detection of organ involvement and closer monitoring of disease progression. Moreover, the introduction of enzyme replacement therapy within the last two decades has changed the natural history of FD as follows: a) increased life expectancy; b) improved morbidity; c) modification of the main cause of morbidity and mortality from renal (kidney) to cardiovascular (heart) events, including heart failure, abnormal heart rhythms, stroke and sudden death. Although symptoms such as palpitations and blackouts are extremely common, information on the frequency of proven abnormal heart rhythms is limited. In addition, the rate and appropriateness of implantation of life-saving devices is very variable, including pacemakers to boost the heart when too slow and cardio-defibrillators that stop the heart when too fast. The main markers of risk in similar diseases such as hypertrophic cardiomyopathy cannot be used in FD. While patients are routinely followed up in clinic with heart tracings and echocardiography (ultrasound of the heart), a recent small study has emphasised that these tests under-estimate the burden of abnormal heart rhythms in patients with advanced FD. The use of continuous heart monitoring with an implantable loop recorder (ILR) has led to a significant change in treatment in 13 out of 15 of FD patients. The investigators believe that more frequent use of ILRs will identify a greater need for change in therapy in many more patients than currently treated, with the aim of reducing morbidity and mortality in this patient cohort. In addition this will provide valuable data to inform an estimate of future risk for these patients.

DETAILED DESCRIPTION:
This is a 3-year open-label multicentre randomised controlled trial assessing arrhythmia burden in patients with Fabry cardiac disease. This is an observational study, but with implantable loop recorder (ILR) insertion at recruitment and removal at end of trial for the intervention arm.

Null hypothesis: There will be no difference in the identification of arrhythmia between patients following standard care compared to patients following standard care but with the addition of ILR monitoring.

Beyond the proposed hypothesis, data collected will be used to inform whether ILR in FD will:

1. Reveal a high burden of unrecognised arrhythmia
2. Lead to frequent treatment modification (anti-coagulation, pacemaker and ICD implantation, ablation)
3. Enable the development of FD specific risk prediction algorithms
4. Identify predictive power of new (Troponin, BNP, lysoGB3, T1 and T2 mapping) and traditional biomarkers

ELIGIBILITY:
Inclusion Criteria:

* Patients with genotypically or enzymatically confirmed FD
* Adults > 18 years of age
* Evidence of cardiac involvement from FD involving either:
* Any ECG abnormality associated with FD
* Low T1 on CMR (below centre-specific normal range according to sex)
* LVH on transthoracic echo (defined as MWT >12mm)

Exclusion Criteria:

* Patient with an existing cardiac device (PPM, ICD or ILR).
* Known dual pathology:
* Known coronary artery disease (positive non-invasive imaging, confirmed myocardial infarction, percutaneous or surgical revascularisation). Patients >40 years old with symptoms that could be from coronary artery disease will have this excluded
* Known cardiomyopathy disease causing mutation (e.g. SCN5, MYBPC3)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2019-09-18 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
First occurrence of atrial fibrillation (AF) requiring anticoagulation | Total monitoring time period in study - 3 years
  This will include all descriptions of AF, which can be defined as:
  1. paroxysmal - self-terminating episodes lasting between 48 hours to 7 days
  2. persistent - intermittent episodes lasting between 7 days to 1 year
  3. permanent - episodes lasting longer than 1 year
First occurrence of bradyarrhythmia requiring cardiac pacing | Total monitoring time period in study - 3 years
  This would include:
  1. Symptomatic significant AV block.
  2. Mobitz type 2 AV block or complete heart block irrespective of symptoms.
First occurrence of supraventricular arrhythmia requiring drug treatment or ablation. | Total monitoring time period in study - 3 years
First occurrence of non-sustained ventricular tachyarrhythmia requiring drug treatment, ICD implantation or ablation | Total monitoring time period in study - 3 years
  This is classified as three or more ventricular beats at a rate >120bpm, for a duration of less than 30 seconds.

SECONDARY OUTCOMES:
Frequency of arrhythmia in patients with and without late gadolinium enhancement (LGE) | 3 years
  The study will aim at quantifying the extent of LGE deposited with myocardial tissue on cardiac MRI scanning. This will subsequently be correlated with the burden of arrhythmia detected to assess for potential risk factors.
Frequency of arrhythmia according to location of myocardial fibrosis (inferolateral vs. non-inferolateral) | 3 years
  The study will aim to correlate the location of myocardial fibrosis with the presence or absence of cardiac arrhythmia to define location of fibrosis as a potential risk factor for arrhythmia.
Frequency of arrhythmia in those patients with a QRS duration greater or less than 120ms | 3 years
Frequency of arrhythmia in those with an atrial size above or below indexed normal range for age and sex | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Richard Steeds, MD, Principal Investigator — University Hospital Birmingham NHS Foundation Trust
Locations (7):
- University of Sydney, Sydney, Australia
- United Kingdom (6):
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham, West Midlands
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - Cardiff and Vale University Health Board, Cardiff
  - Royal Free NHS Foundation Trust, London
  - Salford Royal NHS Foundation Trust, Manchester
  - Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers. Data analysis conducted using anonymised patient data will be shared through publications.

REFERENCES:
- [Derived] Vijapurapu R, Kozor R, Hughes DA, Woolfson P, Jovanovic A, Deegan P, Rusk R, Figtree GA, Tchan M, Whalley D, Kotecha D, Leyva F, Moon J, Geberhiwot T, Steeds RP. A randomised controlled trial evaluating arrhythmia burden, risk of sudden cardiac death and stroke in patients with Fabry disease: the role of implantable loop recorders (RaILRoAD) compared with current standard practice. Trials. 2019 May 31;20(1):314. doi: 10.1186/s13063-019-3425-1. PMID 31151481